CLINICAL TRIAL: NCT00089401
Title: A Phase II Trial Of Isolated Hepatic Perfusion (IHP) With Melphalan For Subjects With Metastatic Unresectable Colorectal Cancers Of The Liver With Disease Refractory To First Line Systemic Chemotherapy
Brief Title: Isolated Hepatic Perfusion With Melphalan in Treating Patients With Unresectable Colorectal Cancer That Has Metastasized to the Liver
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 040229; 04-C-0229; CDR0000378323; NCT00086697 (obsolete NCT alias)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Melphalan

INTERVENTIONS:
Drug: isolated perfusion
Drug: melphalan
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as melphalan, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs in different ways may kill more tumor cells.

PURPOSE: This phase II trial is studying how well isolated hepatic perfusion with melphalan works in treating patients with unresectable colorectal cancer that has metastasized to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response and duration of response in patients with unresectable colorectal cancer metastatic to the liver and refractory to first-line systemic chemotherapy treated with isolated hepatic perfusion with melphalan.

Secondary

* Determine the pattern of recurrence (liver vs systemic) in patients treated with this regimen.
* Determine hepatic progression-free and overall survival in patients treated with this regimen.
* Determine the time to hepatic and systemic progression in patients treated with this regimen.
* Determine quality of life (QOL) in patients treated with this regimen.
* Correlate baseline QOL with length of survival in patients treated with this regimen.

OUTLINE: Patients undergo a limited laparotomy to determine if extrahepatic disease that was not visualized during preoperative scanning is present. Patients found to have peritoneal seeding or unresectable extrahepatic metastatic disease not previously visualized on scans do not receive isolated hepatic perfusion (IHP). Remaining patients undergo IHP with melphalan and hyperthermia therapy. Liver perfusion continues for 1 hour.

Quality of life is assessed at baseline, 6 weeks, and then every 3-4 months for 3 years.

Patients are followed at 6 weeks, every 3-4 months for 3 years, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal cancer

  * Metastatic disease limited to the parenchyma of the liver

    * Patients with limited sites of extrahepatic disease AND who have dominant life-limiting disease in the liver are considered eligible provided the extrahepatic sites can be treated with local ablative measures (e.g., resection or external beam radiotherapy)
    * No other evidence of unresectable extrahepatic disease by radiological studies
* Unresectable hepatic disease defined by > 3 sites of disease in the liver, bilobar disease, or tumor abutting major vascular or ductal structures making anatomic resection with liver function preservation impossible
* Measurable disease
* Refractory to prior first-line systemic chemotherapy

  * Disease progression during or after completion of treatment with an irinotecan- or oxaliplatin-containing regimen for established hepatic metastases

    * Treatment failure is defined as disease progression evidenced by tumor growth OR new lesions on imaging modalities OR increasing carcinoembryonic antigen (CEA)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Hematocrit > 27.0%
* Platelet count > 100,000/mm^3
* WBC > 3,000/mm^3

Hepatic

* Bilirubin < 2.0 mg/dL
* PT ≤ 2 seconds of the upper limit of normal
* ALT and AST elevations secondary to metastatic disease allowed
* Chronic active hepatitis B or C allowed provided there is no evidence of cirrhosis on pathology, radiologic studies, or physical exam
* No history of veno-occlusive disease
* No biopsy proven cirrhosis
* No evidence of significant portal hypertension manifested by ascites, esophageal varices on endoscopy, or radiologic studies showing significant collateral vessels around the organs drained by the portal venous system
* No other liver condition that would preclude study therapy

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* LVEF ≥ 40%
* No ischemic cardiac disease
* No history of congestive heart failure

Pulmonary

* Chronic obstructive pulmonary disease or other chronic pulmonary disease allowed provided pulmonary function test ≥ 50% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* No active infection
* Weight > 30 kg

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy for the malignancy and recovered

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy for the malignancy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy for the malignancy and recovered

Surgery

* See Disease Characteristics

Other

* No concurrent immunosuppressive drugs
* No concurrent chronic anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-07; Primary Completion 2006-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Response
Duration of response

SECONDARY OUTCOMES:
Patterns of tumor recurrence (liver vs systemic)
Progression-free survival
Overall survival
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Libutti, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States